CLINICAL TRIAL: NCT03037060
Title: Exploring Regulation and Function of Dopamine D3 Receptors in Alcohol Use Disorders: A [11C]-(+)-PHNO Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, Principal Investigator, MD, PhD, CCFP, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 052/2016
Record Dates: First submitted 2017-01-16; First posted 2017-01-31 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol use, problem
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Magnetic Resonance Spectroscopy; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): 5 experimental sessions per participant:
  (1) [11C]-(+)-PHNO PET scan, (2), Alcohol Self-Administration, (3) Craving Task, (4) MRI scan and (5) Neuropsychological Assessment.
  Interventions: Other: [11C]-(+)-PHNO PET scan; Other: Alcohol Self-Administration; Other: Craving Task; Other: MRI scan; Other: Neuropsychological Assessment

INTERVENTIONS:
Other: [11C]-(+)-PHNO PET scan — PET scan
Other: Alcohol Self-Administration — Session for assessing motivation for consuming alcohol.
Other: Craving Task — Cue exposure paradigm
Other: MRI scan — MRI scan scan to analyze the PET data will be administered.
Other: Neuropsychological Assessment — Cognitive questionnaires administered over course of study.

SUMMARY:
There is a need to better understand the mechanisms underlying alcohol use and dependence in order to advance the clinical treatment of alcohol dependence. Here, the investigators will use Positron Emission Tomography to determine if there is an up-regulation of D3 receptors in the brains of subjects with alcohol use disorders. The investigators will also investigate the relationship between D3 binding and major phenotypes associated with alcohol use disorders, namely: alcohol cue induced craving and motivation to self-administer alcohol in the laboratory.

DETAILED DESCRIPTION:
Alcohol dependence is a devastating illness with social and medical costs estimated to be 180 billion dollars annually in the US. In the clinical treatment of alcoholism, reducing alcohol consumption in heavy drinkers is a major clinical challenge. As such, there has been much emphasis in both clinical and preclinical research to identify the substrates that mediate craving, excessive drinking and addiction. Identifying the neurobiological mechanisms of alcohol dependence may lead to the development of new and better treatment strategies. Preclinical studies indicate that the D3 receptor is involved in alcohol-cue response and in the motivation to drink alcohol. However, there is currently no data available in human subjects exploring the relationship between D3 and those behavioral responses in subjects with alcohol use disorders.

Aim #1: To measure the [11C]-(+)-PHNO PET binding levels in the brains of subjects with alcohol use disorders.

Aim #2: To determine the relationship between D3 receptor binding and alcohol cue induced craving and motivation to self-administer alcohol in the laboratory.

To achieve designated goals, the investigators will recruit 25 male and female subjects who are non-treatment seekers. After a period of abstinence from alcohol, participants will come to the Centre for Addiction of Mental Health for a [11C]-(+)-PHNO PET scan. Participants will also have additional sessions during which other alcohol-related measures will be assessed (i.e. alcohol cue induced craving and motivation to self-administer alcohol in the laboratory).

ELIGIBILITY:
Inclusion Criteria:

* Subjects will meet diagnostic criteria for alcohol use disorder (mild through severe).
* Willing to abstain from drugs and alcohol prior to study visits
* A negative urine screen for illicit psychoactive drug use
* Willing and capable to provide written informed consent
* Willing to participate in cue exposure and intravenous alcohol administration sessions
* Male and female adults (at least 19 years old)

Exclusion Criteria:

* DSM diagnosis of drug dependence other than alcohol
* Any severe Axis I disorder aside from alcohol use disorder
* Any medical condition requiring immediate investigation
* History of seizures, past or current neurological illness or serious head trauma
* Suicidal ideation
* Pregnancy tested by urine or blood screen or lactation
* Current past or anticipated exposure to radiation exceeding permissible limits as set by the CAMH PET Centre
* Metal implants or paramagnetic objects within the body which may interfere with the MRI
* Claustrophobia or a history of panic attacks
* Any other problem that, in the investigators' opinion, would preclude participation in trial (i.e., complicated withdrawal).
* Currently seeking treatment or attempting to reduce/quit drinking
* History of negative responses to venipuncture procedures (e.g., fainting/vasovagal response)
* Medications or medical disorders for which alcohol consumption is contraindicated

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Dopamine D2/D3 receptor occupancy | One PET scan after 2-7 days of abstinence from alcohol; ~2 hours in duration.
  Dopamine D2/D3 receptor occupancy in the brains of individuals with Alcohol Use Disorders will be quantified using [11C]-(+)-PHNO Positron Emission Tomography (PET). [11C]-(+)-PHNO binding levels will be used to infer receptor occupancy.

SECONDARY OUTCOMES:
Alcohol craving ratings | Cue paradigm session is expected to take ~1 hour and will occur on the PET day.
  Participants' ratings for alcohol craving acquired during the validated Cue-Induced Craving Paradigm (using the Alcohol Urge Questionnaire: 8 items on a 11-point Likert scale) will be correlated to dopamine receptor occupancy (outcome 1).
Effort to obtain alcohol | Single self-administration session will occur on its own day with a time commitment of ~6 hours.
  Laboratory alcohol self-administration paradigm in which participants press a button to intravenously self-administer small doses of alcohol will be used to assess amount of effort expended to obtain alcohol ("break point"). The # of button presses required to obtain the alcohol will increase as per the Progressive Ratio schedule. Regression analysis between effort and [11C]-(+)-PHNO binding (outcome 1) will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre. — http://www.camh.net/research